CLINICAL TRIAL: NCT05321407
Title: Vaccine-induced SARS-CoV-2-specific T Cell Responses in Patients With Primary Immune Deficiency Disease
Brief Title: COVID-19 Vaccine Responses in PIDD Subjects
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Jeffrey Modell Foundation (Unknown); University of North Carolina, Chapel Hill (Other); University of South Florida (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00108422; R21AI168980 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-04-11 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-03

CONDITIONS: X-linked Agammaglobulinemia; XLA; Primary Immune Deficiency; CVID; Common Variable Immunodeficiency; Primary Antibody Deficiencies; Secondary Hypogammaglobulinemia
Keywords: X-linked Agammaglobulinemia; Primary Immune Deficiency; Common Variable Immunodeficiency; SARS CoV 2 Infection; Primary Antibody Deficiencies; COVID-19; Secondary Hypogammaglobulinemia
MeSH Terms: conditions — Bruton type agammaglobulinemia; Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- X-linked agammaglobulinemia (XLA): This study is a non-randomized observational cohort study of participants with XLA who have either received, as standard care, the Pfizer BioNTech BNT162b2 mRNA vaccine or the Moderna mRNA-1273 vaccine. In this protocol, vaccination is entirely voluntary and vaccines are not provided by the study.

SUMMARY:
The goal of our study is to assess the cellular immune responses of participants with antibody deficiency disease before and after immunization with SARS-CoV-2 mRNA vaccines.

DETAILED DESCRIPTION:
Individuals with primary and secondary antibody immunodeficiency are at higher risk for severe COVID-19 disease. Humoral immunity is thought to be the predominant protection against COVID-19, however mRNA vaccines have been shown to elicit both antibody and cellular responses.

The goal of our study is to assess the cellular immune responses of participants with antibody deficiency diseases, including X-linked agammaglobulinemia (XLA), common variable immunodeficiency (CVID), and secondary hypogammaglobulinemia, before and after immunization with SARS-CoV-2 mRNA vaccines.

Our aim is to examine SARS-CoV-2 spike-specific T cell immune responses before and after immunization with mRNA vaccines in a cohort of individuals with antibody deficiencies compared to healthy volunteers. Our secondary objectives include (1) detecting cellular immune response differences between immunized and infected participants, (2) observing cellular immune responses over time, and (3) comparing clinical outcomes between vaccination, infection, and underlying antibody deficiency. The results will show whether antibody deficiency individuals can mount T cell responses to SARS-CoV-2 vaccination or infection, data that are expected to inform health policy of SARS-CoV-2 implementation in immunocompromised individuals. Findings will further provide foundation for larger cohort studies of SARS-CoV-2 vaccination in other immunocompromised populations.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of antibody deficiency with confirmatory lab or genetic testing
2. Stable on immunoglobulin replacement therapy
3. Age >6 months and able to provide consent, or assent with parental consent if <18 years
4. Willing and able to receive the Pfizer BioNTech BNT162b2 mRNA or the Moderna mRNA-1273 vaccines

Exclusion Criteria:

(1) History of other chronic disease with depressed immune function or immune suppressive medication

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 50 subjects with primary antibody deficiency diseases and 50 healthy controls will be enrolled through the Duke University Medical Center's Allergy and Immunology clinics for the Departments of Medicine and Pediatrics, in addition to collaboration with University of North Carolina, Chapel Hill and University of South Florida.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Spike (S) protein-specific T cell responses to stimulation with SARS-CoV-2 wild-type peptides (measured as a percentage of total T cells). | 2 years
Spike (S) protein-specific T cell responses to stimulation with SARS-CoV-2 alpha variant peptides (measured as a percentage of total T cells). | 2 years
Spike (S) protein-specific T cell responses to stimulation with SARS-CoV-2 beta variant peptides (measured as a percentage of total T cells). | 2 years
Spike (S) protein-specific T cell responses to stimulation with SARS-CoV-2 delta variant peptides (measured as a percentage of total T cells). | 2 years
Spike (S) protein-specific T cell responses to stimulation with SARS-CoV-2 omicron variant peptides (measured as a percentage of total T cells). | 2 years

SECONDARY OUTCOMES:
S-specific T cell responses (as a percentage of total T cells) to SARS-CoV-2 vaccination in primary antibody deficiency over time. | 2 years
S-specific T cell responses (as a percentage of total T cells) to SARS-CoV-2 vaccination in secondary antibody deficiency over time. | 2 years
S-specific T cell responses (as a percentage of total T cells) to SARS-CoV-2 in infected participants. | 2 years
S-specific T cell responses (as a percentage of total T cells) to SARS-CoV-2 in vaccinated participants. | 2 years
Number of vaccinated participants who develop severe COVID-19 clinical outcomes. | 2 years
Number of infected participants who develop severe COVID-19 clinical outcomes. | 2 years
Number of antibody deficiency participants who develop severe COVID-19 clinical outcomes. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Sleasman, MD, Principal Investigator — Duke University; Kristina De Paris, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - University of South Florida, St. Petersburg, Florida
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes